CLINICAL TRIAL: NCT07397884
Title: Evaluation of Bone Destruction and Oxidative Stress Markers in Saliva and Peri-implant Sulcus Fluid in Peri-implantitis
Brief Title: Markers of Bone Destruction and Oxidative Stress in Peri-implantitis
Status: Not yet recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Gülbahar Ustaoğlu, Professor, Saglik Bilimleri Universitesi
Other Study IDs: 2025-403
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Periodontal Diseases; Periimplant Diseases
Keywords: Periodontal Diseases; periimplant diseases; Oxidative Stress; Alveolar Bone Loss
MeSH Terms: conditions — Periodontal Diseases; Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Peri-implantitis Group: Patients with at least one dental implant in function for at least 1 year, showing signs of inflammation (BOP/suppuration), probing depth (PD) ≥ 5 mm, and radiographic bone loss ≥ 2 mm.
- Periodontitis Group: Patients with at least one tooth having clinical probing depth ≥ 4 mm, presence of bleeding on probing (BOP), and evidence of radiographic alveolar bone loss.
- Peri-implant Health Group: Patients with implants in function for at least 1 year, showing no signs of inflammation (no BOP), probing depth ≤ 3 mm, and no radiographic bone loss.
- Periodontal Health Group: Systemically healthy individuals with clinical probing depths ≤ 3 mm, minimal plaque and bleeding scores, and no radiographic evidence of bone loss.

SUMMARY:
The aim of this study is to evaluate and compare the levels of bone resorption (RANKL, OPG) and oxidative stress (Nitrotyrosine, NQO1) markers, along with pro-inflammatory cytokines (IL-1β), in the saliva and peri-implant sulcular fluid (PISF) of patients with peri-implantitis, periodontitis, and healthy individuals. The study seeks to determine the diagnostic value of these biomarkers in the early detection and progression of peri-implant diseases.

DETAILED DESCRIPTION:
Patients applying to the University of Health Sciences, Gulhane Faculty of Dentistry, Department of Periodontology, will be screened according to the inclusion and exclusion criteria. Following clinical and radiographic examinations, participants will be categorized into four groups (n=20 per group): Periodontitis, Peri-implantitis, Periodontal Health, and Peri-implant Health. All clinical parameters, including Plaque Index (PI), Gingival Index (GI), Bleeding on Probing (BOP), Probing Depth (PD), and Clinical Attachment Loss (CAL), will be recorded at six sites per tooth/implant using a Williams periodontal probe.

The biological sample collection protocol will be conducted as follows:

Saliva Collection: To minimize circadian rhythm variations, unstimulated whole saliva samples (3 ml) will be collected between 9:00 AM and 10:00 AM. Patients will be instructed to refrain from eating, drinking, or oral hygiene procedures for at least one hour prior to collection. Samples will be centrifuged at 1,000g for 10 minutes to remove cellular debris, and the supernatant will be stored at -80°C until laboratory analysis.

Peri-implant Sulcular Fluid (PISF) and Gingival Crevicular Fluid (GCF) Collection: Samples will be obtained from the site with the deepest probing depth in each participant. The area will be isolated with cotton rolls and gently dried with an air syringe to prevent salivary contamination. Periopaper strips will be inserted into the sulcus/pocket for 30 seconds. Strips contaminated with blood or visible saliva will be discarded.

Laboratory Analysis: The concentrations of Interleukin-1 beta (IL-1β), Nitrotyrosine, Receptor Activator of Nuclear Factor Kappa-B Ligand (RANKL), Osteoprotegerin (OPG), and NAD(P)H: Quinone Oxidoreductase 1 (NQO1) will be quantified in both saliva and PISF/GCF samples using commercially available Enzyme-Linked Immunosorbent Assay (ELISA) kits according to the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy volunteers aged 18-65. For Peri-implantitis group: Implants in function for ≥1 year, radiographic bone loss ≥ 2 mm, probing depth (PD) ≥ 5 mm, and presence of bleeding on probing (BOP) or suppuration.

For Periodontitis group: At least one tooth with PD ≥ 4 mm, presence of BOP, and radiographic bone loss.For Healthy groups: PD ≤ 3 mm, no clinical inflammation (BOP-), and no radiographic bone loss.

(According to the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases) -

Exclusion Criteria:Presence of systemic diseases (e.g., diabetes, rheumatoid arthritis, osteoporosis).

Use of antibiotics, anti-inflammatory, or immunosuppressive drugs within the last 3 months.

Pregnancy or breastfeeding.

Smoking (current smokers).

History of periodontal or peri-implant surgical treatment within the last 6 months.

Implant failure (mobility).

Signs of acute infection (fever, systemic symptoms).

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who apply to the University of Health Sciences, Gulhane Faculty of Dentistry, Department of Periodontology, and meet the specific clinical and radiographic criteria for peri-implantitis, periodontitis, or health.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Salivary and Peri-implant Sulcular Fluid (PISF) IL-1β Levels. | At the baseline clinical examination (Day 0).
  The concentration of Interleukin-1 beta (IL-1β), a pro-inflammatory cytokine, will be measured in picograms per milliliter (pg/mL) using ELISA kits to evaluate the severity of inflammation and bone destruction.

SECONDARY OUTCOMES:
Salivary and Peri-implant Sulcular Fluid (PISF) Nitrotyrosine Levels | Baseline (at the time of clinical examination)
  Concentration of Nitrotyrosine will be measured in saliva and PISF samples using ELISA kits. Nitrotyrosine serves as a biochemical marker of nitrosative stress to evaluate oxidative damage.
Salivary and Peri-implant Sulcular Fluid (PISF) NQO1 Levels | Baseline (at the time of clinical examination)
  NAD(P)H: Quinone Oxidoreductase 1 (NQO1) levels will be measured using ELISA kits to assess the local and systemic antioxidant defense response.
Salivary and Peri-implant Sulcular Fluid (PISF) RANKL Levels | Baseline (at the time of clinical examination)
  Receptor Activator of Nuclear Factor Kappa-B Ligand (RANKL) levels will be measured to evaluate osteoclast activation and bone destruction potential.
Salivary and Peri-implant Sulcular Fluid (PISF) OPG Levels | Baseline (at the time of clinical examination)
  Osteoprotegerin (OPG) levels will be measured. OPG acts as a decoy receptor for RANKL, and its level indicates the body's attempt to inhibit bone resorption.
Clinical Attachment Loss (CAL) and Probing Depth (PD) | Baseline (at the time of clinical examination)
  CAL and PD will be measured in millimeters (mm) at six sites per tooth/implant using a Williams periodontal probe to assess the severity of tissue destruction.
Plaque Index (PI) and Gingival Index (GI) | Baseline (at the time of clinical examination)
  PI and GI will be recorded using Silness-Löe and Löe-Silness indices (scored 0-3) to evaluate oral hygiene status and gingival inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Gülbahar Ustaoğlu, Professor, Principal Investigator — University of Health Sciences, Gulhane Faculty of Dentistry, Department of Periodontology

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared to protect participant privacy.